CLINICAL TRIAL: NCT05244876
Title: Effect of Back School-based Intervention on Non-specific Neck Pain in Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Pablo Hernandez-Lucas, Associate professor in health sciences, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 931919
Record Dates: First submitted 2022-01-21; First posted 2022-02-17 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Neck Pain; Exercise Therapy; Health Education
MeSH Terms: conditions — Neck Pain; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The person analysing the data does not know which group he or she belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Intervention based on the Back School was carried out for 8 weeks with a frequency of two sessions per week, with a total of 16 sessions lasting 45 min.
  Interventions: Behavioral: Back school
- Control group (No Intervention): I declare that I will not change my lifestyle during the study process.

INTERVENTIONS:
Behavioral: Back school — Intervention was carried out for 8 weeks with a frequency of two sessions per week, with a total of 16 sessions lasting 45 min. Of all the sessions, 14 had a practical focus and the other two had a theoretical focus. In the practical part, strengthening and stretching exercises were performed. In the theoretical part, self-management and pain neuroscience education were performed.
  Arms: Experimental group

SUMMARY:
The study consists of a theoretical and practical intervention based on the Back School. This intervention will be carried out over 8 weeks with a frequency of two sessions per week, for a total of 16 sessions of 45 minutes duration. Of all the sessions, 14 had a practical focus (strength and stretching exercises) and the other two had a theoretical focus (self-management techniques and pain neuroscience education). In addition, they had an initial session and a session at the end of the of the intervention in which measurements of the different variables were taken (The Visual Analogue Scale; Neck Disability Index; Tampa Scale Of kinesiophobia).These variables will be measured on two occasions, at the beginning of the study and at the end of the intervention, an average of 2 months.

The clinical practice guidelines highlight the importance of neck pain prevention through exercise an education. There are previous studies of the effects of theoretical and practical programmes based on back school on the lumbar region but not on the cervical region. Therefore, the aim of this study is to investigate the effects of a BS-based intervention on neck pain and functionality as well as kinesiophobia and quality of life in adults. The hypothesis previously hypothesised that this BS-based intervention would have positive effects on pain, functionality, kinesiophobia and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age.
* With non-specific neck pain for at least three months, with pain intensity (30-70 on a VAS).

Exclusion Criteria:

* Any previous neck or shoulder surgery, fibromyalgia, cervical radiculopathy/myelopathy, history of the whiplash injury, cognitive disorder.
* Missing more than two Back School sessions.
* Not being able to attend the measurement sessions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Through study completion, an average of 2 months.
  The visual analog scale (VAS) is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge (=VAS score).
Neck Disability Index | Through study completion, an average of 2 months.
  The NDI can be scored as a raw scorer doubled and expressed as a percent. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. Points summed to a total score. The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage.
Short-Form Health Survey-36 | Through study completion, an average of 2 months.
  Short-Form Health Survey (SF-36) was used to measure quality of life.The SF-36 explores people's physical and mental health. It consists of 36 items that assessed eight dimensions of health status: social function, physical function, emotional role, physical role, mental health, vitality, physical pain, and general health. Scores ranged from 0 (worst health status) to 100 (best health status).
Tampa Scale Of Kinesiophobia. | Through study completion, an average of 2 months.
  This scale measures kinesiophobia. The total scale score ranges from 11 to 44, where 11 means no kinesiophobia and 44 means severe kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Pablo Hernández Lucas, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hernandez-Lucas P, Leiros-Rodriguez R, Lopez-Barreiro J, Garcia-Soidan JL. Effects of back school-based intervention on non-specific neck pain in adults: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2023 Apr 17;15(1):60. doi: 10.1186/s13102-023-00666-8. PMID 37069599